CLINICAL TRIAL: NCT00067288
Title: Meaning-Centered Psychotherapy in Advanced Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: R21AT001031-01 (NIH); Breitbart
Record Dates: First submitted 2003-08-14; First posted 2003-08-15 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Lymphoma, Non-Hodgkin; Neoplasms
Keywords: Stage 3 cancer;; Stage 4 cancer;; solid tumor cancer;; Non-Hodgkin's Lymphoma;; solid tumors;; end-stage cancer;; group psychotherapy;; psychotherapy;; emotional support;; support groups
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms

INTERVENTIONS:
Behavioral: Meaning-Centered Group Psychotherapy
Behavioral: Standard Supportive Group Psychotherapy

SUMMARY:
We have developed an 8-week Meaning-Centered Group Psychotherapy designed to help patients with advanced cancer sustain or enhance a sense of meaning, peace and purpose despite the limitations of their cancer illness. This project's overall aim is to explore the feasibility and efficacy of this new and unique psychotherapy intervention for advanced cancer patients in enhancing psychological and spiritual well-being and quality of life by comparing it with a standard supportive group psychotherapy.

DETAILED DESCRIPTION:
As per Brief Summary

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older;
* English speaking;
* Stage III or IV solid-tumor or Non-Hodgkin's Lymphoma;
* Receiving ambulatory care at Memorial Sloan-Kettering Cancer Center in New York City;

Exclusion Criteria:

* Significant psychiatric disturbance sufficient, in the investigator's judgment, to preclude participation in a group-format intervention;
* Presence of cognitive impairment disorder, such as delirium or dementia that is sufficient, in the investigator's opinion, to preclude meaningful participation and/or informed consent;
* Karnofsky Performance Rating Scale below 50 or physical limitations or illness severity sufficient to preclude participation in outpatient group psychotherapy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118
Dates: Start 2002-05; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: William Breitbart, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Christopher Gibson, PhD — Project Coordinator Memorial Sloan-Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Institute for Cancer Research, New York, New York, United States